CLINICAL TRIAL: NCT01273480
Title: An Open-Label, Multicenter Study to Assess the Potential Effects of Rifampin on the Pharmacokinetics of Trabectedin in Subjects With Advanced Malignancies
Brief Title: A Study to Assess the Potential Effects of Rifampin on the Pharmacokinetics of Trabectedin in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017536; ET743OVC1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-12-23; First posted 2011-01-10 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Neoplasm Metastases
Keywords: Trabectedin, YONDELIS; Rifampin (RIFADIN); Antineoplastic Agents; Solid tumors; Locally advanced or metastatic disease; Chemotherapy; Pharmacokinetics
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 002 (Experimental): Sequence 2 Cycle 1: Trabectedin 1.3 mg/m2 i.v. on Day 1 followed by 2 rifampin 300 mg capsules once daily on Days 24-28 followed by Cycle 2 2 rifampin capsules prior to trabectedin 1.3 mg/m2 i.v. on Day 1 of Cycle 2. Dexamethasone 20 mg i.v. administered prior to trabectedin in each cycle.
  Interventions: Drug: Sequence 1; Drug: Sequence 2
- 001 (Experimental): Sequence 1 Cycle 1: 2 rifampin 300 mg capsules 1x daily for 5 days followed by 2 rifampin capsules prior to trabectedin 1.3 mg/m2 i.v. on Day 1 followed 28 days later by cycle 2 trabectedin 1.3 mg/m2 i.v. on Day 1. Dexamethasone 20 mg i.v. administered prior to trabectedin in each cycle.
  Interventions: Drug: Sequence 2; Drug: Sequence 1

INTERVENTIONS:
Drug: Sequence 1 — Cycle 1: 2 rifampin 300 mg capsules 1x daily for 5 days followed by 2 rifampin capsules prior to trabectedin 1.3 mg/m2 i.v. on Day 1 followed 28 days later by cycle 2 trabectedin 1.3 mg/m2 i.v. on Day 1. Dexamethasone 20 mg i.v. administered prior to trabectedin in each cycle.
  Arms: 002
Drug: Sequence 2 — Cycle 1: Trabectedin 1.3 mg/m2 i.v. on Day 1 followed by 2 rifampin 300 mg capsules once daily on Days 24-28 followed by Cycle 2, 2 rifampin capsules prior to trabectedin 1.3 mg/m2 i.v. on Day 1 of Cycle 2. Dexamethasone 20 mg i.v. administered prior to trabectedin in each cycle.
  Arms: 001
Drug: Sequence 1 — Cycle 1: 2 rifampin 300 mg capsules 1x daily for 5 days followed by 2 rifampin capsules prior to trabectedin 1.3 mg/m2 i.v. on Day 1 followed 28 days later by cycle 2 trabectedin 1.3 mg/m2 i.v. on Day 1. Dexamethasone 20 mg i.v. administered prior to trabectedin in each cycle.
  Arms: 001
Drug: Sequence 2 — Cycle 1: Trabectedin 1.3 mg/m2 i.v. on Day 1 followed by 2 rifampin 300 mg capsules once daily on Days 24-28 followed by Cycle 2, 2 rifampin capsules prior to trabectedin 1.3 mg/m2 i.v. on Day 1 of Cycle 2. Dexamethasone 20 mg i.v. administered prior to trabectedin in each cycle.
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the potential effects of rifampin on blood levels of trabectedin after administration to patients with advanced malignancies.

DETAILED DESCRIPTION:
This is an open-label study (patients will know the names of the study drugs they receive), randomized (patients will be assigned 1 of 2 treatment sequences by chance) that is designed to examine the pharmacokinetics (blood levels) and to assess survival and safety of trabectedin when coadministered with rifampin in patients with advanced malignancies. Study drugs include trabectedin and rifampin. Trabectedin is a drug being developed to treat patients with cancer that will be administered intravenously (i.v.) through a catheter (tube) into a central vein over a period of 3 hours once every 28 days with and without rifampin. Rifampin is an antibiotic that may interfere with the action of trabectedin that will be taken orally (by mouth) as capsules. In addition, dexamethasone, a drug used to prevent nausea and vomiting in chemotherapy patients that may have protective effects on the liver, will be administered to patients before the administration of trabectedin. In the study, 3 patients will initially be randomized sequentially to Treatment Sequence 1 or Treatment Sequence 2 to evaluate safety. If the safety and pharmacokinetic data collected from these 3 patients is deemed acceptable, additional patients will be randomized to 1 of 2 treatment sequences. Patients who complete the treatment phase of the study or who are discontinued due to rifampin toxicity, and who in the opinion of the investigator would derive an overall clinical benefit from further treatment with trabectedin, will have the opportunity to continue treatment with trabectedin in the optional extension phase. The dose and schedule of trabectedin may be modified by the treating physician in the optional extension phase to be more appropriate for the type of malignancy being treated. Patients will receive 20 mg of i.v. dexamethasone (or its equivalent) prior to trabectedin administration in all cycles. Patients randomized to Sequence 1 will receive rifampin 600mg 1X daily(6 doses)+trabectedin 1.3 mg/m2 i.v. followed 28 days later by trabectedin 1.3 mg/m2 i.v. Patients randomized to Sequence 2 will receive trabectedin 1.3 mg/m2 i.v. followed 28 days later by rifampin 600mg 1X daily(6 doses)+trabectedin 1.3mg/m2 i.v. Dexamethasone 20 mg i.v., or equivalent will be administered 30 minutes prior to trabectedin administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic disease, any solid tumor except hepatocellular carcinoma, who have relapsed or had progressive disease following standard of care treatment with chemotherapy prior to enrollment, or intolerant to prior standard of care treatment with chemotherapy
* Patients with Eastern Cooperative Oncology Group (ECOG) score of <=2
* Patients able to receive dexamethasone
* Patients with hepatic function variables: total bilirubin <=upper limit of normal (ULN), alkaline phosphatase (ALP) <=1.5 ULN and liver function test results (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) of <=2.5x ULN

Exclusion Criteria:

* Patients with previous exposure to trabectedin
* Patients with cancer that has metastasized (spread) to the central nervous system
* Patients with known liver disease
* Patients who had a myocardial infarct (heart attack) within 6 months before enrollment or who have any other clinically significant or unstable medical condition as assessed by the Investigator
* Patients unable to have a central catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of trabectedin | At protocol-specified time points up to 8 days during each 28-day cycle in Sequence 1 and up to 6 days during each 28-day cycle in Sequence 2
Pharmacokinetics of rifampin | 1 day during Sequence 1 and Sequence 2 after rifampin is coadministered with trabectedin

SECONDARY OUTCOMES:
Number of patients with adverse events | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin
Findings from clinical laboratory evaluations | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin
Findings from vital signs measurements | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin
Findings from physical examinations | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Philadelphia, Pennsylvania
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Machiels JP, Staddon A, Herremans C, Keung C, Bernard A, Phelps C, Khokhar NZ, Knoblauch R, Parekh TV, Dirix L, Sharma S. Impact of cytochrome P450 3A4 inducer and inhibitor on the pharmacokinetics of trabectedin in patients with advanced malignancies: open-label, multicenter studies. Cancer Chemother Pharmacol. 2014 Oct;74(4):729-37. doi: 10.1007/s00280-014-2554-1. Epub 2014 Aug 7. PMID 25100135
- See also: An Open-Label, Multicenter Study to Assess the Potential Effects of Rifampin on the Pharmacokinetics of Trabectedin in Subjects With Advanced Malignancies — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=870&filename=CR017536_CSR.pdf